CLINICAL TRIAL: NCT06629974
Title: The Effects of an Empowerment Program for Parents of Children With Autism: A Randomised Controlled Trial
Brief Title: The Effects of an Empowerment Program for Parents of Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCBU-SBF-RK-01
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Autism; Parenting; Motivational Interviewing
Keywords: Autism; Parent training; Empowerment; Parental self-efficacy; Parental stress; Care burden
MeSH Terms: conditions — Autistic Disorder; Empowerment; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: This unblinded, randomized controlled interventional study with two parallel groups involved parents of children diagnosed with autism. Participants were stratified according to their educational status, and each participant was assigned a number. Participants within each stratum were assigned to either the intervention or control groups using simple randomization with a table of random numbers.The study was completed with a total of 69 participants: 34 in the intervention group and 35 in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this group were administered the pre-intervention introductory information form, The Parental Self-Efficacy Scale, the Zarit Care Burden Scale, the Perceived Stress Scale and the Family Empowerment Scale. Then, a group empowerment training program consisting of four sessions in total was applied to the participants. Two motivational interview sessions were conducted with each participant in the intervention group 10 days after the empowerment training program. One month after the motivational interview sessions were completed, post-test data were collected.
  Interventions: Behavioral: Parental empowerment program
- Control group (No Intervention): No intervention was applied to the control group. The data collection tools applied to the intervention group in the pre-test and post-test were also applied to the control group.

INTERVENTIONS:
Behavioral: Parental empowerment program — The empowerment program consisted of two parts: the empowerment training program for parents and motivational interviews.
  The empowerment training program was prepared to enable parents to carry out the care process more effectively in areas where parents have difficulties caring for their children with autism. Within the scope of the empowerment training program, parents were trained on the importance of play and communication, problems and management in the field of nutrition, sleep problems and management, safety and protection from accidents, and problems and management in the field of self-care.
  Ten days after the empowerment training program, two face-to-face motivational interviews were conducted with each participant in the intervention group. Each participant had a one-week break between the first and second motivational interviews. Each motivational interview session lasted approximately 25-30 minutes.
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the effectiveness of an empowerment program that includes both parent training and motivational interviewing for parents of children with autism, supporting their competence in the care of their children.

DETAILED DESCRIPTION:
This study was conducted to evaluate the effectiveness of an empowerment program for parents of children with autism to support their competence in caring for their children. This randomized controlled study was conducted in Manisa city center/Turkey, in 2022. A total of 69 parents (intervention: 34, control: 35) were included in this unblinded, two-group randomized controlled interventional study. A parent empowerment program, including four parental training sessions and two motivational interview sessions, were applied to the parents in the intervention group. The Parental Self-Efficacy Scale, Zarit Care Burden Scale, Perceived Stress Scale, and Family Empowerment Scale were used to evaluate the effectiveness of the empowerment program.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were having a child diagnosed with ASD between the ages of 6 and 14, being literate, and volunteering to participate in the study.

Exclusion Criteria:

* Having a child with a concomitant disability or disease (e.g., epilepsy, attention deficit, and hyperactivity disorder, other physical or mental disabilities), previous participation in an education program with similar content, or parents who did not participate in at least two-thirds of the empowerment training program or did not attend all motivational interview sessions were excluded from the study, and their data were not included in the analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
The parental self-efficacy scale scores | Three months
  The scale was developed by Guimond et al. (2005) to measure the self-efficacy of parents of children with disabilities regarding parenting skills (Guimond et al., 2005). The Turkish adaptation of the scale was first made by Diken (2007) and then by Cavkaytar et al. (2014) (Cavkaytar et al., 2014; Diken, 2007). The Parental Self-Efficacy Scale is a seven-point Likert-type rating scale consisting of 17 items. The lowest and highest values that can be taken from the scale are 17 and 119. Higher scores indicate higher self-efficacy perceptions. The Cronbach Alpha internal consistency coefficient value of the scale was calculated as 0.95 (Cavkaytar et al., 2014). The Cronbach's Alpha internal consistency coefficient value of the scale in this study is 0.96.
The zarit care burden scale scores | Three months
  The Zarit Care Burden Scale was developed by Zarit et al. in 1980 and adapted to Turkish by Inci and Erdem (2006). The scale is a 22-item, five-point Likert-type scale used to evaluate the stress experienced by caregivers of individuals in need of care. A minimum score of 0 and a maximum score of 88 can be obtained from the scale. The higher the score obtained from the scale, the higher the care burden felt. The Cronbach's Alpha internal consistency coefficient value of the scale was found to be 0.75 in the original study (Inci and Erdem, 2006; Zarit et al., 1980) and 0.89 in this study.
The perceived stress scale scores | Three months
  The Perceived Stress Scale was developed by Cohen et al. (1983) and adapted into Turkish by Eskin et al. This 14-item, five-point Likert-type scale has two sub-dimensions: inadequate self-efficacy perception and stress/discomfort perception. Higher scores indicate higher levels of perceived stress. The Cronbach's alpha internal consistency coefficient for the entire scale was 0.90, with the sub-dimensions scoring 0.86 and 0.83, respectively (Cohen et al., 1983; Eskin et al., 2013). In this study, the Cronbach's alpha internal consistency coefficient was found to be 0.75 for the overall scale and 0.73 and 0.75 for the sub-dimensions, respectively.
The family empowerment scale scores | Three months
  The Family Empowerment Scale, developed by Singh et al. (1995) and adapted into Turkish by Karakul et al. (2018), consists of 34 questions and three sub-dimensions, rated on a four-point Likert scale. Higher scores indicate stronger family empowerment. The Cronbach's alpha internal consistency coefficient for the entire scale was 0.89. The sub-dimensions had the following Cronbach's alpha values: 0.79 for the Family subdimension, 0.83 for the Service system subdimension, and 0.79 for the Community/Political sub-dimension (Karakul et al., 2018; Singh et al., 1995). In this study, Cronbach's alpha coefficient was 0.79 for the overall scale, 0,83 for the family dimension, 0,89 for the services sub-dimension and 0,85 the community/political sub-dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Damla Şahin Büyük, Phd, Principal Investigator — Manisa Celal Bayar University
Locations (1):
- Manisa Celal Bayar University, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data may be shared with individual researchers upon request after the study has been completed and published; however, for data security reasons, sharing the data prior to publication is not being considered.

REFERENCES:
- [Background] Karakul, A., Akgül, E. A., Doğan, P., Sarı, H. Y., 2018. Psychometric properties of the family empowerment scale in Turkish. Izmir Katip Celebi Univ. J. Health Sci. 3(3) 111.
- [Background] Singh, N. N., Curtis, W. J., Ellis, C. R., Nicholson, M. W., Villani, T. M., Wechsler, H. A., 1995. Psychometric analysis of the family empowerment scale. J. Emotion. Behav. Disord. 3, 85-91.
- [Background] Eskin, M., Harlak, H., Demirkıran, F., Dereboy, Ç., 2013. Adaptation of the perceived stress scale into Turkish: reliability and validity analysis. New Symp. J. 51, 132-140.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Inci, F., Erdem, M., 2006. Adaptation of the Caregiving Burden Scale into Turkish, its validity and reliability. Anatol. J. Nurs. Health Sci. 11, 85-95.
- [Background] Guimond, A., Moore, H., Aier, D., Maxon, E., Diken, I., 2005. Parental self-efficacy instrument for children with disabilities (PSICD): Short version. Unpublished scale. Arizona: Arizona State University.
- [Background] Diken, I. H., 2007.Turkish mothers' self-efficacy beliefs and styles of interactions with their children with language delays. Early Child Dev. Care 179, 425-436.
- [Background] Cavkaytar, A., Aksoy, V., & Ardıç, A., 2014. Updating the validity and reliability study of the parent self-efficacy scale. Anadolu J. Educ. Sci. Int. 4, 69-76.
- [Result] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Derived] Sahin Buyuk D, Ozmen D. Effectiveness of a Parent Empowerment Program for Parents of Children with Autism: A Randomized Controlled Trial. Child Care Health Dev. 2025 Sep;51(5):e70148. doi: 10.1111/cch.70148. PMID 40751565